CLINICAL TRIAL: NCT02229721
Title: Female Sexual Dysfunction in the Menopause: Effect of Intranasal Oxytocin Administration on Sexual Function and Activity
Brief Title: Effect of Chronic Intranasal Oxytocin Administration on Sexual Function in Pre- and Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Dana Muin, Univ. Prof. Michaela Bayerle-Eder, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-001310-34
Record Dates: First submitted 2014-08-27; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Female Sexual Dysfunction
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Syntocinon Nasalspray 32 IU (Active Comparator): Over 8 weeks, intranasal oxytocin (32 IE) or placebo will be self-administered by women prior to sexual intercourse. Following a washout period of 2 weeks, a cross-over will take place and patients switched to the alternate group for another 8 weeks.
  The recommended dose is four puffs per nostril, containing 32 IU of synthetic oxytocin, administered up to 50 minutes prior to sexual activity. The maximal dose should not exceed four puffs per nostril per day; the minimum dose was twice weekly.
  Interventions: Drug: Syntocinon Nasalspray; Drug: Placebo Nasalspray
- Placebo Nasalspray (Placebo Comparator): Over 8 weeks, intranasal oxytocin (32 IE) or placebo will be self-administered by women prior to sexual intercourse. Following a washout period of 2 weeks, a cross-over will take place and patients switched to the alternate group for another 8 weeks.
  The recommended dose is four puffs per nostril, administered up to 50 minutes prior to sexual activity. The maximal dose should not exceed four puffs per nostril per day; the minimum dose was twice weekly.
  Interventions: Drug: Syntocinon Nasalspray; Drug: Placebo Nasalspray

INTERVENTIONS:
Drug: Syntocinon Nasalspray — Over 8 weeks, intranasal oxytocin (32 IE) or placebo will be self-administered by women prior to sexual intercourse. Following a washout period of 2 weeks, a cross-over will take place and patients switched to the alternate group for another 8 weeks.
  The recommended dose is four puffs per nostril, containing 32 IU of synthetic oxytocin, administered up to 50 minutes prior to sexual activity. The maximal dose should not exceed four puffs per nostril per day; the minimum dose was twice weekly.
  Other Names: Oxytocin
Drug: Placebo Nasalspray — Over 8 weeks, intranasal oxytocin (32 IE) or placebo will be self-administered by women prior to sexual intercourse. Following a washout period of 2 weeks, a cross-over will take place and patients switched to the alternate group for another 8 weeks.
  The recommended dose is four puffs per nostril, administered up to 50 minutes prior to sexual activity. The maximal dose should not exceed four puffs per nostril per day; the minimum dose was twice weekly.

SUMMARY:
The purpose of this study is to determine whether intranasal oxytocin is effective in comparison to placebo in improving female sexual dysfunction in pre- and postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to attempt sexual intercourse and/ or masturbation at least two times per week
* Ongoing relationship for at least 3 months
* Female subjects aging 40 years and more, Male subjects must be older than 18
* The participation in this study should be of free choice to male partners
* Willingness to perform a pregnancy test every month (for pre-menopausal subjects)
* Willingness to use contraception during the study period (for pre-menopausal subjects)
* Normal findings in the urogenital tract unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Primary sexual dysfunction
* sexual abuse
* severe psychiatric diseases
* untreated conditions and medication intake with associated reduction of sexual function.
* In male partners: any severe andrological or related medical problem.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function | 22 weeks
  Assessment by standardized questionnaires including Female Sexual Function Index (FSFI), Female Sexual Distress Scale (FSDS), Sexual Quality of Life-Female (SQOL-F), Sexual Activity Record (SAR), and Sexual Interest and Desire Inventory-Female (SIDI-F).

SECONDARY OUTCOMES:
Hamilton Depression Scale (HDS) | 22 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Muin DA, Sheikh Rezaei S, Tremmel-Scheinost M, Salama M, Luger A, Wolzt M, Husslein PW, Bayerle-Eder M. Men's sexual response to female partner's intranasal oxytocin administration for hypoactive sexual desire disorder: an open prospective cohort study. Fertil Steril. 2017 Mar;107(3):781-787.e3. doi: 10.1016/j.fertnstert.2016.12.003. Epub 2017 Feb 8. PMID 28189292
- [Derived] Muin DA, Wolzt M, Marculescu R, Sheikh Rezaei S, Salama M, Fuchs C, Luger A, Bragagna E, Litschauer B, Bayerle-Eder M. Effect of long-term intranasal oxytocin on sexual dysfunction in premenopausal and postmenopausal women: a randomized trial. Fertil Steril. 2015 Sep;104(3):715-23.e4. doi: 10.1016/j.fertnstert.2015.06.010. Epub 2015 Jul 4. PMID 26151620